CLINICAL TRIAL: NCT02252536
Title: Randomized, Double Blind, Placebo-Controlled Trial of the Safety and Efficacy of HORIZANT (Gabapentin Enacarbil) Extended-Release Tablets for the Treatment of Alcohol Use Disorder
Brief Title: HORIZANT (Gabapentin Enacarbil Extended-Release Tablets) for the Treatment of Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCIG - 006
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; alcoholism; alcohol dependence; drinking alcohol
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Matching placebo, sugar pill
  Interventions: Drug: Placebo
- Gabapentin Enacarbil (Active Comparator): 600 mg Gabapentin Enacarbil (Horizant)
  Interventions: Drug: gabapentin enacarbil

INTERVENTIONS:
Drug: gabapentin enacarbil — Horizant Extended Release Tablets, 600 mg, white to off-white, oval shaped tablets, taken 2 times per day
  Other Names: Horizant Extended Release Tablets
  Arms: Gabapentin Enacarbil
Drug: Placebo — Placebo tablet, white to off-white, oval shaped tablets, taken 2 times per day
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to determine whether gabapentin enacarbil is effective in the treatment of problems with alcohol.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet each one of the following inclusion criteria in order to be eligible for participation in the study:

1. Be at least 21 years of age.
2. Have a current (past 12 months) DSM-5 diagnosis of AUD.
3. Have a BAC by breathalyzer equal to 0.000 when s/he signed the informed consent document (either just prior to or immediately after signing consent).
4. Be seeking treatment for problems with alcohol.

Additional will be evaluated in clinic.

Exclusion Criteria:

Evaluations will be conducted in clinic.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Z. Litten, Ph.D., Study Chair — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (10):
- United States (10):
  - University of California Los Angeles, Los Angeles, California
  - Friends Research Institute, San Francisco, California
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Mount Sinai St. Luke's Hospital, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a Phase 2, randomized, double-blind, placebo controlled, parallel-group 26-week treatment clinical trial. Candidates responded by telephone to advertisements at 10 academic sites in the US between June 2015 and February 2017.
Period: Overall Study
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Started | 173 | 173
Completed | 168 | 170
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Gabapentin Enacarbil | Total
Number analyzed (Participants) | 168 | 170 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.4) | 50.7 (10.3) | 50.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 48 | 115
  Male | 101 | 122 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 14 | 32
  Not Hispanic or Latino | 146 | 150 | 296
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 35 | 63
  White | 126 | 117 | 243
  More than one race | 10 | 9 | 19
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 168 | 170 | 338

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With no Heavy Drinking Days (PSNHDD)
Description: The primary objective of the study is to compare the efficacy of HORIZANT (gabapentin enacarbil) Extended-Release Tablets 600 mg twice daily (BID) with matched placebo on the primary alcohol consumption outcome endpoint, percentage of subjects with no heavy drinking days (PSNHDD) during the last 4 weeks of treatment, among patients with Alcohol Use Disorder (AUD).
Time Frame: Weeks 22-25
Measure: Number; unit: percentage of subjects with NHDD
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
percentage of subjects with NHDD | 17.3 | 24.1

2. Secondary Outcome: Percentage of Subjects Abstinent From Alcohol (Key Secondary Endpoint)
Description: Timeline Follow-back drinking data is used to calculate the % of subjects that report not drinking alcohol during weeks 22-25
Time Frame: Weeks 22-25
Population: no imputation was performed so the number analyzed is reduced
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 136 | 146
Participants | 16 | 17

3. Secondary Outcome: Percentage of Subjects With a World Health Organization (WHO) Drinking Risk Category Decrease of at Least 1-level
Description: Timeline Follow Back data is used to calculate the % of participants that decrease at least 1-level WHO drinking risk category. The WHO has developed a drinking risk categorical scale that can be used in a responder analysis approach to assess clinically relevant decreases in alcohol consumption (Aubin et al-2015). The WHO 1- and 2-level decrease endpoints are the percentage of subjects experiencing at least 1- and 2-level decrease in WHO levels of alcohol consumption, respectively, from the level at baseline (the period including the 28 days before screening) to the level during the last 4 weeks of the maintenance phase (Study Weeks 22-25). The WHO levels are as follows:
  Males Females Low Risk 1 to 40g 1 to 20g Medium Risk 41 to 60g 21 to 40g High Risk 61 to 100g 41 to 60g Very High Risk 101+g 61+g
Time Frame: Weeks 22-25
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 134 | 146
Participants | 107 | 115

4. Secondary Outcome: Percentage of Subjects With a World Health Organization (WHO) Drinking Risk Category Decrease of at Least 2-levels
Description: as for outcome 3
Time Frame: Weeks 22-25
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 134 | 146
Participants | 69 | 80

5. Secondary Outcome: Percentage of Days Abstinent Per Week
Description: Timeline Follow Back daily drinking data used to calculate the % of days abstinent per week.
Time Frame: Weeks 22-25
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
percentage of days | 49 (3.9) | 49.3 (3.9)

6. Secondary Outcome: Percentage of Heavy Drinking Days Per Week
Description: Timeline Follow Back data used to calculate the % of heavy drinking days per week. Heavy drinking is 4+ drinks per day for females and 5+ drinks per day for males
Time Frame: Weeks 22-25
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
percentage of days | 46.5 (4.2) | 43.1 (4.1)

7. Secondary Outcome: Weekly Mean Number of Drinks Per Week
Description: Timeline Follow Back data used to calculate the weekly mean number of drinks per week
Time Frame: Weeks 22-25
Measure: Least Squares Mean (Standard Error); unit: drinks per week
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
drinks per week | 21.4 (2.4) | 23.1 (2.3)

8. Secondary Outcome: Weekly Mean Drinks Per Drinking Day
Description: Timeline Follow Back daily drinking data used to calculate the weekly mean drinks per drinking day
Time Frame: Weeks 22-25
Measure: Least Squares Mean (Standard Error); unit: drinks per drinking day
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
drinks per drinking day | 3.9 (0.4) | 4.1 (0.4)

9. Secondary Outcome: Cigarettes Per Week Among Smokers
Description: A quantity frequency interview of three questions to assess cigarette smoking behavior and other tobacco/nicotine containing products use during the study: 1) "Over the past week, on how many days did you smoke cigarettes?", 2) "On the days you smoked during the past week, how many cigarettes did you smoke on average?", and 3) "Have you used any other tobacco or nicotine containing products besides cigarettes in the past week (e.g., cigars, cigarellos, pipes, bidis, or smokeless tobacco such as pan, chewing tobacco, or snuff, or nicotine replacement therapies such as patch or gum)?".
Time Frame: Weeks 22-25
Measure: Least Squares Mean (Standard Error); unit: cigarettes per week
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
cigarettes per week | 61.4 (8.3) | 71 (8.3)

10. Secondary Outcome: Alcohol Craving Score [Alcohol Craving Scale - Short Form (ACQ-SR-R)]
Description: The ACQ-SR-R contains 12-items adapted from the 47-item ACQ-NOW developed by Singleton et al (1994) to assess craving for alcohol among alcohol users in the current context (right now). Each item has a 1 to 7 raw score (from strongly disagree to strongly agree). Items 3, 8, and 11 are reverse keyed. A general craving index is derived by summing all items and dividing by 12. Minimum score is 1 and maximum score is 7. Higher scores are indicative of higher craving.
  Mixed effects models as stated in Section 9.4.3 of the SAP will be generated for the total score and for the 4 subscales. Covariates for these models will be identified
Time Frame: Weeks 24 and 26
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
scores on a scale | 2.5 (0.1) | 2.5 (0.1)

11. Secondary Outcome: Alcohol Related Consequences (ImBIBe) Score
Description: ImBIBe is a 15-item questionnaire in which the subject responds on a 5-point scale (0-4) responses to questions on the consequences of alcohol use. This scale was adapted from the Drinker Inventory of Consequences questionnaire based on FDA recommendations on patient reported outcomes (Miller & Tonigen-1995). The potential range is 0-60. A higher score indicates a worse outcome. The questions are added together. A question that is missing is imputed with the average value of all other questions in the questionnaire.The total score is the sum of the individual item scores.
  Mixed effects models as stated in Section 9.4.3 will be generated for the total score. Covariates for these models will be identified
Time Frame: Weeks 24 and 26
Measure: Least Squares Mean (Standard Error); unit: total score
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
total score | 8.3 (0.7) | 9.6 (0.7)

12. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI) Score
Description: The PSQI is a 19-item questionnaire assessing the subject's overall sleep experience in the past 30 days (Buysse et al-1989). The lower the overall score, the better the person sleeps. The tool has an adequate internal reliability, validity and consistency for clinical and community samples of the various populations. Range is (0-21); >6 indicative of "poor" sleep quality.
Time Frame: Week 26
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
score | 4.4 (0.2) | 4.9 (0.2)

13. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: The BAI consists of 21 questions about how the subject has been feeling in the last week, expressed as common symptoms of anxiety (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). This inventory was designed to minimize the overlap with depression scales (Beck et al-1988).The BAI has a maximum score of 63. The standardized cutoffs for anxiety severity are: 0-7: minimal level of anxiety 8-15: mild anxiety 16-25: moderate anxiety 26-63: severe anxiety
Time Frame: Week 26
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
score | 3.3 (0.5) | 4.6 (0.4)

14. Secondary Outcome: Beck Depression Inventory - II
Description: The BDI-II is a 21-item multiple choice questionnaire that is used for measuring the severity of depression (Beck et al-1966). Each item is scored on a scale value of 0 to 3. The standardized cutoffs for depression severity are:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression
Time Frame: Week 26
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Sugar Pill | Gabapentin Enacarbil
Number analyzed (Participants) | 168 | 170
score | 5.2 (0.5) | 6.5 (0.5)

ADVERSE EVENTS:
Time Frame: AEs were assessed from Week 1 - Week 29.
Description: General symptoms were collected via an open ended question: "How have you been feeling since your last visit or the last time we spoke?"
Arm/Group | Sugar Pill | Gabapentin Enacarbil
All-Cause Mortality (participants affected / at risk) | 0/168 | 1/170
Serious Adverse Events (participants affected / at risk) | 6/168 | 8/170
Other Adverse Events (participants affected / at risk) | 155/168 | 157/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=168) | Gabapentin Enacarbil (N=170)
Alcohol Withdrawal (Nervous system disorders) | 0 (0) | 3 (3)
migraine with left eye drooping (Nervous system disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Orbital Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Laceration complicated by orbital fracture (Infections and infestations) | 0 (0) | 1 (1)
Acute Intoxication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bradycardia during colonoscopy (Cardiac disorders) | 1 (1) | 0 (0)
Suicidality (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Stomach Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcohol Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Comminuted impacted fracture of the right humeral head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=168) | Gabapentin Enacarbil (N=170)
Diarrhea (Gastrointestinal disorders) | 10 | 11
Nausea (Gastrointestinal disorders) | 23 | 17
Blood Pressure diastolic increased (Investigations) | 42 | 43
Headache (Nervous system disorders) | 47 | 38
Fatigue (General disorders) | 26 | 44
Blood Pressure Systolic increase (Investigations) | 32 | 33
Dizziness (Nervous system disorders) | 23 | 36
Aspartate Aminotransferase Increased (Investigations) | 26 | 24
Gamma-glutamyltransferase increased (Investigations) | 19 | 30
Somnolence (Nervous system disorders) | 16 | 30
Nasopharyngitis (Infections and infestations) | 21 | 19
Upper respiratory tract infection (Infections and infestations) | 17 | 22
Insomnia (Nervous system disorders) | 17 | 18
Alanine aminotransferase increased (Investigations) | 19 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 19 | 11
Vomiting (Gastrointestinal disorders) | 8 | 15
Blood creatinine increased (Investigations) | 8 | 14
Anxiety (Psychiatric disorders) | 7 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 5
Blood bilirubin increased (Investigations) | 9 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Paraesthesia (Nervous system disorders) | 6 | 11
Abnormal dreams (Psychiatric disorders) | 9 | 6
Rash (Skin and subcutaneous tissue disorders) | 13 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 3
Agitation (Psychiatric disorders) | 3 | 9
Depressed mood (Psychiatric disorders) | 9 | 3
Tremor (Nervous system disorders) | 1 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restricts disclosure until the main study paper is published.

DOCUMENTS (2):
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT02252536/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02252536/SAP_001.pdf